CLINICAL TRIAL: NCT04650139
Title: Coronary Interventions Ulm - Coronary Chronic Total Occlusions
Acronym: CSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Ulm (Other)
Responsible Party: Principal Investigator, Bruno Correia, Investigator, University Hospital Ulm
Other Study IDs: 0925-0586
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Chronic Total Occlusion
MeSH Terms: interventions — Percutaneous Coronary Intervention; Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- successful CTO
  Interventions: Procedure: PCI - percutaneous coronary intervention
- non- successful CTO
  Interventions: Procedure: PCI - percutaneous coronary intervention

INTERVENTIONS:
Procedure: PCI - percutaneous coronary intervention — percutaneous coronary intervention
  Other Names: drug eluting stents, Scaffolds, drug eluting ballons

SUMMARY:
The aim of the proposed project is to provide the long-term results after a recanalization attempt of chronically occluded coronary arteries.

To investigate recanalization attempt of chronically occluded coronary arteries at the Ulm University Hospital. As shown, it is known that successful recanalization of a chronic occlusion is associated with a lower event rate (reduced mortality and the need for operative myocardial revascularization) compared to unsuccessful recanalization (drug therapy). The standard in the therapy of successfully recanalized chronic occlusions is the use of drug-releasing vascular supports.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years

Coronary intervention in chronic coronary artery occlusion

Occlusion > 3 months

Indication for PTCA or recanalization according to guidlines

such as:

Symptoms of the patient

Evidence of myocardial ischemia (stress ECG, scintigraphic

Methods, magnetic resonance imaging, stress echocardiography)

pathological intracoronary flow reserve, prognostic

Exclusion Criteria:

* No chronic occlusion,
* Contraindication to anti-platelet therapy

Acetylsalicylic acid plus clopidogrel for at least 3 months such as e.g.

with florid gastrointestinal ulcer disease,

History of hemorrhagic stroke

or urgent non-postponable surgical intervention.

Basic disease with a life expectancy of less than 12 months (here as a rule

no indication for PTCA or reopening available)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with CTO
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
MACE | 1 year
  major adverse cardiac event

SECONDARY OUTCOMES:
TLR | 1 year
  target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- University Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided